CLINICAL TRIAL: NCT04471480
Title: Paclitaxel and Carboplatin Plus PD-1 Inhibitors Combined With Anlotinib for Advanced Esophageal Cancer(ESCC)
Brief Title: TC Plus PD-1 Inhibitors Combined With Anlotinib for Advanced Advanced Esophageal Cancer
Acronym: TC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dong Wang (Other)
Responsible Party: Sponsor-Investigator, Dong Wang, Head of Oncology, Third Military Medical University
Organization: Third Military Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCAC-ESCC-01
Record Dates: First submitted 2020-07-12; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: ESCC
Keywords: PD-1; anlotinib
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A，TCCA (Experimental): paclitaxel for Injection 175 mg/m2,IV, d1/paclitaxel for Injection (Albumin Bound) 260mg/m2,IV, d1, q3w +carboplatin AUC 4-6,IV, d12,q3w +anlotinib 10mg, PO, d1-14, q3w +camrelizumab 200 mg, IV, d1, q3w, after the treatment for 4-6 cycles, camrelizumab plus anlotinib for maintenance therapy until PD or intolerable toxicity
  Interventions: Drug: TC/PD-1 inhibitor/anlotinib
- group B，TCC (Experimental): paclitaxel for Injection 175 mg/m2,IV, d1/paclitaxel for Injection (Albumin Bound) 260mg/m2,IV, d1, q3w +carboplatin AUC 4-6,IV, d12,q3w +camrelizumab 200 mg, IV, d1, q3w, after the treatment for 4-6 cycles, camrelizumab for maintenance therapy until PD or intolerable toxicity
  Interventions: Drug: TC/PD-1 inhibitor/anlotinib
- group C，TC (Other): paclitaxel for Injection 175 mg/m2,IV, d1/paclitaxel for Injection (Albumin Bound) 260mg/m2,IV, d1, q3w +carboplatin AUC 4-6,IV, d12,q3w
  Interventions: Drug: TC/PD-1 inhibitor/anlotinib

INTERVENTIONS:
Drug: TC/PD-1 inhibitor/anlotinib — chemotherapy and immunotherapy plus antiangiogenic therapy
  Other Names: TC/PD-1 inhibitor

SUMMARY:
A Controlled Clinical Study of TC/PD-1 Inhibitors Combined With anlotinib as First-line Treatment for Advanced ESCC

DETAILED DESCRIPTION:
The incidence rate of esophageal cancer is high in China and mainly squamous cell carcinoma. In recent years, although the level of surgery, radiotherapy and chemotherapy of esophageal cancer has improved, and studies have confirmed the role of anlotinib and PD-1 mAb in the posterior line treatment of esophageal squamous cell carcinoma, the prognosis of esophageal cancer is still not ideal. How to expand the clinical benefits of immunotherapy in esophageal cancer has become a research hotspot. Recent studies have shown that PD-1 mAb combined with other therapies with different mechanisms can improve the efficacy of immunotherapy. In the impawer150 study, platinum containing dual drug chemotherapy plus anti angiogenesis therapy combined with immunotherapy showed statistically and clinically significant PFS benefits in the first-line treatment of advanced non-small-cell lung cancer, which provides a new choice for the first-line treatment of advanced non-small-cell lung cancer. So far, there is no report on the first-line treatment of advanced esophageal squamous cell carcinoma with platinum containing dual drug chemotherapy plus anti angiogenesis drugs combined with immunotherapy. The purpose of this study is to evaluate the efficacy of cisplatin plus cisplatin in the treatment of advanced esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in the study and signed the informed consent;
2. Age 18-75, both male and female;
3. Histologically or cytologically confirmed advanced or metastatic (stage IIIB, III C or IV) ESCC .
4. At least one measurable lesion according to RECIST 1.1,which should not be treated locally, such as radiotherapy.
5. ECOG PS 0-1- Page 3 of 5 [DRAFT] -
6. Expected survival ≥ 3 months
7. Patients who never received systemic therapy in the past, including radiotherapy ,chemotherapy, targeted therapy and immunotherapy , or patients who relapsed more than 6 months after adjuvant chemotherapy.
8. The main organ functions accorded with the following criteria within 7 days before treatment:

(1)Blood routine examination ( without blood transfusion in 14 days): hemoglobin (HB) ≥ 90 g/L; neutrophil absolute value (ANC) ≥ 1.5 *109/L; platelet (PLT) ≥80 *109/L.

(2) Biochemical tests should meet the following criteria: 1) total bilirubin (TBIL) ≤1.5 times of upper limit of normal (ULN); 2) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 *ULN, if accompanied by liver metastasis, ALT and AST ≤ 5* ULN; 3) serum creatinine (Cr) ≤ 1.5* ULN or creatinine clearance rate (CCr) ≥ 60 ml/min;4) Serum albumin (≥35g/L). (3) Doppler echocardiography: left ventricular ejection fraction (LVEF) ≥the low limit of normal value (50%).

9 Tissue samples should be provided for biomarker analysis (such as PD-L1 ) Patients who could not provide new tissues could provide 5-8 paraffin sections of 3-5 μm by archival preservation.

Exclusion Criteria:

1. Severe allergic reactions to humanized antibodies or fusion proteins in the past
2. known to have hypersensitivity to any component contained in Endostar or antibody preparations;
3. Diagnosed of immunodeficiency or received systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 14 days before the study, allowing physiological doses of glucocorticoids (≤10mg/day prednisone or equivalent);
4. Patients with active, known or suspected autoimmune diseases. Patients with type I diabetes, hypothyroidism requiring hormone replacement therapy, skin disorders requiring no systemic treatment(such as vitiligo, psoriasis or alopecia). Patients who would not triggers can be included.
5. Serious heart disease, include congestive heart failure, uncontrollable high-risk arrhythmia, unstable angina pectoris, myocardial infarction, and severe valvular disease.
6. Patients treated targeted drugs such as bevacizumab, sunitinib, sorafenib, imatinib, famitinib, regiffenil, apatinib and anlotinib
7. Patients recieved systemic antineoplastic therapy, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or mitomycin C within 6 weeks before the grouping),recieved over-extended-field radiotherapy (EF-RT) within 4 weeks before the grouping or limited-field radiotherapy to evaluate the tumor lesions within 2 weeks before the grouping
8. Positive hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus antibody (HCV Ab), indicating acute or chronic infection.
9. Patients with active pulmonary tuberculosis (TB) infection judged by chest X-ray examination, sputum examination and clinical physical examination. Patients with active pulmonary tuberculosis infection in the previous year should be excluded even if they have been treated; Patients with active pulmonary tuberculosis infection more than a year ago should also be excluded unless the course and type of antituberculosis treatment previously were appropriate.
10. Patients with brain metastases with symptoms or symptoms controlling less than 2 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate(ORR) | approximately 18 months
  complete response(CR)+partial response(PR) according to RECIST 1.1
overall survival (OS) | approximately 36 months
  overall survival is defined as the time from randomization to death from any cause

SECONDARY OUTCOMES:
progression-free survival(PFS) | approximately 36 months
  progression-free survival is defined as the time from enrollment to the date of first document disease progression or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu M, Pu Y, Jiang Y, Liu Y, Feng Y, Zhao X, Li M. Anlotinib plus camrelizumab and chemotherapy as first-line treatment in patients with advanced esophageal squamous cell carcinoma. Sci Rep. 2025 Jul 1;15(1):22275. doi: 10.1038/s41598-025-06625-2. PMID 40595001